CLINICAL TRIAL: NCT01588756
Title: Development of a New Non-radioactive Test for Measuring Glomerular Filtration Rate Using the Tetrapeptide N-acetyl-Ser-Asp-Lys-Pro-amide (AcSDKP-NH2)
Acronym: AcSDKP-NH2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOM08193
Record Dates: First submitted 2012-04-02; First posted 2012-05-01 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Healthy; Chronic Kidney Disease
Keywords: Chronic kidney disease; GFR; Inulin; 51Cr-EDTA; ASDKP-NH2; Healthy male 18-35 yrs old, non smokers, non allergic; Or Male/female 18-80 yrs old with chronic Kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AcSDKP-NH2 inuline (Experimental): AcSDKP-NH2 inuline, Once intravenous administration of 100 µg or less
  Interventions: Drug: AcSDKP-NH2 inuline
- AcSDKP-NH2 Cr-EDTA (Experimental): AcSDKP-NH2 Cr-EDTA, Once intravenous administration of 100 µg or less
  Interventions: Drug: AcSDKP-NH2 Cr-EDTA

INTERVENTIONS:
Drug: AcSDKP-NH2 inuline — Once intravenous administration of 100 µg or less
  Arms: AcSDKP-NH2 inuline
Drug: AcSDKP-NH2 Cr-EDTA — Once intravenous administration of 100 µg or less
  Arms: AcSDKP-NH2 Cr-EDTA

SUMMARY:
The purpose of the study is to validate a new reference marker for evaluation of renal function (glomerular filtration rate).

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a worldwide public health problem with an increasing incidence and prevalence, poor outcomes (kidney failure, complications of decreased kidney function and cardiovascular disease), and high cost. Some of the adverse outcomes can be prevented or delayed by early detection and treatment. However, CKD is frequently underdiagnosed and undertreated. The glomerular filtration rate (GFR) is considered as the best index of renal function. The clinical action plan promoted by International Guidelines groups refers to GFR values. Despite recent improvements, prediction equations developed in order to estimate GFR elicit a huge lack of accuracy when considering the individual patient, especially in case of early CKD. Rigorous assessment of GFR requires the measurement of urinary or plasma clearance of an ideal exogenous filtration marker which is either non-radioactive (inulin, iothalamate, or iohexol) or radioactive ( 51Cr-EDTA or 99mTc DTPA. Measuring clearance with the use of exogenous markers is difficult to perform in clinical practice because it is expensive and cumbersome and needs specialised laboratories and thus, is underused. There is an unmet need for the development of a new non-radioactive GFR tracer that could combine both the analytical accuracy of radioactive tracers and the simplicity of its measurement. Such a tracer should improve clinical care and follow-up of patients.

ELIGIBILITY:
Inclusion Criteria:

* Phase I: 18-35 years male
* Phase I: healthy volunteers
* Phase II: 18-80 years patients (both sex)
* Phase II: with Chronic Kidney Disease

Exclusion Criteria:

* Phase I: Smokers
* Phase I: Allergic

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
glomerular filtration rate | between day 7 and day 21
  NAcSDKP clearance for GFR measurement is compared to inuline and 51Cr-EDTA clearance in two phase I studies in 50 healthy subjects. GFR is first assessed at equilibrium by measuring urinary clearances of inuline and NAcSDKP continuously co-infused after a loading dose; and second by plasma clearances of 51Cr-EDTA and NAcSDKP after a single IV bolus. Optimal conditions for using NAcSDKP as a marker for GFR and the tolerability of the peptide are assessed during these studies. Then, a phase IIa study will be performed to compare the 2 methods in 45 patients with various degrees of renal failure.

SECONDARY OUTCOMES:
safety | One month extended to 3 months safety follow up
  all adverse events (clinical or biological adverse events)

CONTACTS AND LOCATIONS:
Overall Officials: Michel AZIZI, MD, PhD, Principal Investigator — Université Paris-Descartes, Faculté de Médecine; Assistance Publique Hôpitaux de Paris, Hôpital Européen Georges Pompidou, Centre d'Investigations Cliniques; INSERM, CIC 9201, F-75015 Paris, France
Locations (1):
- Clinical Investigation Center, European George Pompidou Hospital, Paris, France

REFERENCES:
- [Result] Mesmin C, Cholet S, Blanchard A, Chambon Y, Azizi M, Ezan E. Mass spectrometric quantification of AcSDKP-NH2 in human plasma and urine and comparison with an immunoassay. Rapid Commun Mass Spectrom. 2012 Jan 30;26(2):163-72. doi: 10.1002/rcm.5326. PMID 22173804